CLINICAL TRIAL: NCT01895998
Title: Quantifying the Presence of Lung Disease and Pulmonary Hypertension in Children With Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00040933
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; pulmonary hypertension; airway hyperreactivity; acute chest syndrome
MeSH Terms: conditions — Anemia, Sickle Cell; Hypertension, Pulmonary; Acute Chest Syndrome | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Albuterol — This medication will be used as routine part of pulmonary function testing to assess for airway hyperreactivity. This is routinely done in a clinical capacity for pediatric patients with various pulmonary disease processes.

SUMMARY:
The proposed research study is a cross-sectional study enrolling young children with sickle cell disease between 5 and 12 years of age. They will be screened as outpatients for consent to perform pulmonary function testing (PFT) and echocardiography. In addition, the degree of bronchodilator response will be assessed at each session. To estimate presence of pulmonary hypertension, echocardiography will be performed at the time of PFT measures.

Study Design:

1. Enroll children aged 5 to 12 years of age with sickle cell disease (HbSS, HbSC, HbS beta plus thalassemia, HbS beta zero thalassemia, and HbS OArab) who are established patients within the Duke Pediatric Sickle Cell Clinic.
2. Perform a chart review of all enrolled subjects to obtain specific details regarding birth history, nutritional status (weight, height), family history, sickle cell genotype, parental smoking history, recent laboratory parameters, parental smoking history, any concurrent conditions (atopy, asthma, airway anomaly), history of sickle cell complications and prescribed medications.
3. Perform spirometry and plethysmography with the administration of albuterol.
4. Before or after completion the PFT session, the patient will have echocardiography in the PFT lab area
5. Using medical record information, determine number of hospitalizations for any pulmonary symptoms indicative of acute chest syndrome (ACS) (dyspnea, fever, wheezing, hypoxia, cough, chest pain). In addition, we will track any respiratory or cardiac symptoms or therapies for each subject 6 years after enrollment up to age 18 years using the registry.
6. As standard of care, refer any child identified as having lung disease or pulmonary hypertension to a pediatric pulmonologist and/or cardiologist for monitoring, treatment and ongoing care.

ELIGIBILITY:
Inclusion Criteria:

* children aged 5 to 12 years of age with sickle cell disease (HbSS, HbSC, HbS beta plus thalassemia, HbS beta zero thalassemia, and HbS OArab)
* established patients within the Duke Pediatric Sickle Cell Clinic.
* Subjects must have been full-term at birth
* any race or gender

Exclusion Criteria:

* significant chromosomal/congenital anomalies
* hemodynamically significant congenital heart disease (arrhythmia requiring medication, defects with chronic hypoxia, single ventricle physiology, heart failure)
* any child within 3 weeks of a respiratory tract infection, an asthma attack, an episode of ACS or of a vaso-occlusive or hemolytic crisis.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Presence of obstructive or restrictive lung disease | One testing session- approximately 3 hours total
  Obstructive lung disease will be defined as forced expiratory volume in 1 second (FEV1), or forced vital capacity (FVC) < 80% predicted based on normative data for age, sex, height, weight and race. Restrictive lung disease will be defined as total lung capacity (TLC) <80% predicted based on normative data for age, sex, height, weight and race.

SECONDARY OUTCOMES:
Presence of pulmonary hypertension | one testing session- approximately 15 minutes
  Pulmonary hypertension will be defined as a tricuspid regurgitation (TR) jet gradient that predicts a pulmonary artery (PA) systolic pressure greater than half of the systemic systolic pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Peterson-Carmichael, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States